CLINICAL TRIAL: NCT02928718
Title: The Association Between Post-ERCP Acute Pancreatitis and Various Genetic Mutations
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hyub Lee, Professor, Seoul National University Hospital
Other Study IDs: 2015-1992
Record Dates: First submitted 2016-07-21; First posted 2016-10-10 (Estimated); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Acute Pancreatitis
Keywords: Post-ERCP pancreatitis; Genetic variation
MeSH Terms: conditions — Pancreatitis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- High risk patients: Patients who are at high risk of post-ERCP pancreatitis, who have at least one of the following factors: clinically suspected sphincter of Oddi dysfunction, history of post-ERCP pancreatitis, pancreatic sphincterotomy, precut sphincterotomy, difficult cannulation, balloon dilatation of intact sphincter, endoscopic ampullectomy, and 2≥minor criteria(an age of less than 50 years and female sex, a history of recurrent pancreatitis (≥2 episodes), three or more injections of contrast agent into the pancreatic duct with at least one injection to the tail of the pancreas, excessive injection of contrast agent into the pancreatic duct resulting in opacification of pancreatic acini,the acquisition of a cytologic specimen from the pancreatic duct with the use of a brush).
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — Two expert endoscopists will perform ERCP. Patients will be sedated with midazolam(2-5mg) and pethidine(25-50mg) with careful monitoring. Duodenoscope (TJF-240 or TJF-260; Olympus Corp., Tokyo, Japan) will be used. Cholangiography or pancreatography will be gathered after selective bile duct or pancreatic duct cannulation. Therapy such as endoscopic sphincterotomy, stent insertion, and etc., will be done.

SUMMARY:
Pancreatitis remains the most common complication of ERCP, with the reported incidence ranging from 2% to 9%. Although 80% of cases are mild, a significant number of patients may develop severe pancreatitis, that means additional morbidity and risk for death. ERCP, despite the development of new diagnostic tools, remains a widely used procedure, so post-ERCP pancreatitis is a problem with significant impact. Several studies and meta-analyses helped us to recognize special factors that put an individual in high risk for the development of post-ERCP pancreatitis. Among these factors special interest presents the history of post-ERCP pancreatitis as an independent risk factor for a new episode of post-ERCP pancreatitis. It seems that some individuals have a genetically predisposed susceptibility in this particular complication. The aim of the present study is to investigate the possible genetic variation associated with post-ERCP pancreatitis using whole genome sequencing.

DETAILED DESCRIPTION:
This study includes patients who are at high risk of post-ERCP pancreatitis. Blood samples will be gathered to investigate the possible genetic variation associated with post-ERCP pancreatitis using whole genome sequencing. DNA for whole genome sequencing will be extracted using DNA extraction kit (Qiagen Inc., Hinden, Germany) and the concentration & purity of DNA will be measured using Nanodrop (Nano Drop Technologies, Wilmington, DE, USA) or fluorometric quantitation(Qubit fluorometer). Genetic variations which are associated with acute pancreatitis will be searched using whole genome sequencing. Post-ERCP pancreatitis is the primary outcome. Medical records and data of genetic variations will be reviewed for identifying possible risk factors and genetic variations associated with post-ERCP pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo ERCP with high risk factors of post-ERCP pancreatitis

Exclusion Criteria:

* <18 years old
* current pancreatitis (<72hrs before ERCP)
* pregnant woman, breast-feeding woman
* patient refusal
* contraindication of ERCP
* patients who would only be treated of bile duct such as a change of stent with previous endoscopic sphincterotomy
* chronic pancreatitis
* patients who underwent gastrectomy (Billroth II or Roux-en Y anastomosis)
* patients who have pancreatic or distal bile duct cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at high risk of post-ERCP pancreatitis, who have at least one of the following factors: clinically suspected sphincter of Oddi dysfunction, history of post-ERCP pancreatitis, pancreatic sphincterotomy, precut sphincterotomy, difficult cannulation, balloon dilatation of intact sphincter, endoscopic ampullectomy, and 2≥minor criteria(an age of less than 50 years and female sex, a history of recurrent pancreatitis (≥2 episodes), three or more injections of contrast agent into the pancreatic duct with at least one injection to the tail of the pancreas, excessive injection of contrast agent into the pancreatic duct resulting in opacification of pancreatic acini,the acquisition of a cytologic specimen from the pancreatic duct with the use of a brush).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Post-ERCP pancreatitis | 24 hours after ERCP
  Clinical pancreatitis, amylase at least 3 x normal >24h after ERCP

SECONDARY OUTCOMES:
Severe post-ERCP pancreatitis | 24 hours after ERCP
  Pancreatitis requiring hospitalization >10 days, intervention(percutaneous drainage or surgery), development of necrosis, or pseudocyst
hyperamylasemia without symptom | 24 hours after ERCP
  amylase at least 3 x normal > 24h after ERCP, no abdominal pain
Length of stay | 3mo
  Duration of hospitalization
Mortality | 3mo
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyub Lee, MD. PhD., Principal Investigator — Department of internal medicine and liver research institute, Seoul national university hospital, Seoul, Korea
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Choi YH, Lim Y, Jang DK, Ahn DW, Ryu JK, Paik WH, Kim YT, Kim JH, Lee SH. Genetic susceptibility to post-endoscopic retrograde cholangiopancreatography pancreatitis identified in propensity score-matched analysis. Korean J Intern Med. 2023 Nov;38(6):854-864. doi: 10.3904/kjim.2022.404. Epub 2023 Oct 23. PMID 37867141